CLINICAL TRIAL: NCT00845793
Title: The Meal Tray as a Tool and Platform to Change Eating Habits Among Hospitalized Diabetic Patients - An Intervention Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Ram Weiss MD PhD, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HMO- 0584-08
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Nutrition; Lifestyle modifications
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Nutritional guidance — The guidance will be performed using the food tray during the hospitalization and will consist of meeting the nutritionist and receiving brochures along with the meal tray focusing on constituents and elements of the diet. The served meals will consist of elements recommended for patients with T2DM (such as whole grains, low fat dairy products and canola oil).

SUMMARY:
This protocol is intended to test whether a focused nutritional intervention in hospitalized patients with type 2 diabetes can have an impact on long term eating habits, physical activity and anthropometric parameters.

The rational is to use the food tray as a means of conveying simple and practical nutritonal and behavioral messages.

DETAILED DESCRIPTION:
Patients hospitalized at Hadassah Medical Center who have type 2 diabetes will relieve a focused nutritional intervention using mainly the food tray during the hospitalization. The intervention will be administered by the hospital nutrition team.

At baseline (upon admission) - medical data will be collected as well as nutritional and behavioral questionnaires will be administered. The intervention will take place during the hospitalization period. Follow up using the same tools will be performed at 3 and 12 month.

We believe that the hospitalization period, even for reasons non related to diabetes, is a window of opportunity to implement lifestyle changes.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-80 years
* Diagnosis of type 2 diabetes
* Speaking and reading Hebrew

Exclusion Criteria:

* Chronic medical condition requiring a specific diet
* Non Hebrew speaking
* Pregnant women

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the results of the nutrition quality questionnaire | 3 and 12 months

SECONDARY OUTCOMES:
Changes in anthropometric measures Changes in physical activity levels | 3 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel